CLINICAL TRIAL: NCT06189209
Title: A Phase II, Multi-center, Single-arm, Open-label Study to Assess the Efficacy and Safety of Tenalisib, a PI3K δ/γ, and SIK3 Inhibitor, in Patients With Metastatic Triple Negative Breast Cancer (TNBC)
Brief Title: Efficacy and Safety of Tenalisib in Patients With Metastatic Triple Negative Breast Cancer (TNBC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Collaborators: Incozen Therapeutics Pvt Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP6530-2301
Record Dates: First submitted 2023-12-08; First posted 2024-01-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Cancer (TNBC)
Keywords: RP6530; Tenalisib
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — tenalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm, Open label study (Experimental): Single agent Tenalisib [RP6530 (PI3k delta, gamma and SIK3 inhibitor)]
  Interventions: Drug: Tenalisib

INTERVENTIONS:
Drug: Tenalisib — Tenalisib will be administered 800mg/ 400mg BID, orally
  Other Names: RP6530

SUMMARY:
This is a Phase II, open-label, single-arm, study, designed to evaluate the efficacy and safety of tenalisib in patients with metastatic TNBC, who have received at least one but not more than 3 prior therapies in a metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have histologically confirmed TNBC.
2. Patients who have received at least 1 but not more than 3 prior chemotherapy regimens in a metastatic setting.
3. Patients with at least one measurable lesion, per RECIST version 1.1 at baseline . Bone-only disease is not permitted.
4. ECOG performance status 0 to 2.
5. Adequate bone marrow, liver, and renal function

Exclusion Criteria:

1. Cancer therapy/ any cancer investigational drug within 3 weeks (21 days) or 5 half-lives (whichever is shorter).
2. Patient who has not recovered from acute toxicities of previous therapy except treatment-related alopecia.
3. Prior exposure to PI3K inhibitors (e.g., alpelisib, buparlisib) for breast cancer.
4. Major surgery within 4 weeks of starting study treatment.
5. Patient with symptomatic uncontrolled brain metastasis.
6. Ongoing immunosuppressive therapy including systemic corticosteroids.
7. History of severe cutaneous reactions.
8. Concurrent disease or condition that would interfere with study participation
9. Pregnancy or lactation.
10. Any severe and/or uncontrolled medical conditions or other conditions that could affect patient participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 1 year
  It is defined as the percentage of patients achieving complete response (CR), partial response (PR), or stable disease (SD) for 16 weeks or longer.
Duration of Clinical Benefit (DoCB) | 1 year
  It is defined as the time from the first dose to disease progression or death on study from any cause, whichever occurs first in patients who achieve CR, PR or SD for 16 weeks or longer.
Overall Response Rate (ORR) | 1 year
  Overall Response is defined as sum of CR and PR.
Progression Free Survival (PFS) | 1 year
  It is defined as the time from the first dose to disease progression or death on study from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events as Assessed by CTCAE v5.0 | 1 year
  Number of adverse events reported by the patients
Trough plasma concentrations of tenalisib/metabolite | 1 year
  plasma concentrations of drug
Correlation of efficacy to baseline mutational status | 1 year
  Baseline mutational status and its correlation with efficacy

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - HCG City Cancer Center, Vijayawada, Andhra Pradesh
  - Narayana Hrudayala Majumdar Shaw Hospital, Bangalore, Karnataka
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Mumbai Oncocare Centre, Mumbai, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Nobel Hospital, Pune, Maharashtra
  - Meenakshi Mission Hospital & Research Center, Madurai, Tamil Nadu
  - Nizams Institute of Medical Science, Hyderabad, Telangana
  - Health Point Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No